CLINICAL TRIAL: NCT00196820
Title: A Multicenter Phase II Study to Determine the Efficacy of Capecitabine as First Line Monochemotherapy in Patients With HER2 Negative, Medium-risk, Metastatic Breast Cancer
Brief Title: Mono Efficacy of Capecitabine (MoniCa)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBG 39; Eudract Number: 2005-000074-51
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2008-05

CONDITIONS: Breast Cancer
Keywords: Metastatic breast cancer; HER2 negative, medium-risk, metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Capecitabine 2000 mg/m2 orally day 1-14 q day 22 until progression, unacceptable toxicity, patient's request or withdrawal from study
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine

SUMMARY:
Study done in patients with metastatic breast cancer in order to determine the efficacy of capecitabine

DETAILED DESCRIPTION:
Study design:

Prospective, open phase II trial

Treatment:

Capecitabine 2000 mg/m² orally day 1-14 q day 22 until progression, unacceptable toxicity, patient's request or withdrawal from study

Primary objective

To determine the time to disease progression in patients with HER2 negative metastatic breast cancer after 1st line monochemotherapy with capecitabine

Secondary objectives

1. To determine the objective response rate
2. To determine the duration of response
3. To determine the clinical benefit defined as CR, PR, or stable disease ≥ 24 weeks
4. To evaluate the safety and toxicity of capecitabine
5. To assess quality of life within 1 year after start of capecitabine treatment
6. To determine overall survival
7. To determine the objective response rate in male patients
8. To evaluate QoL the modified Brunner Score (Appendix 7 )

Tertiary objective

To determine the DPD and Proteomics in serum

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements.
2. Histologically confirmed carcinoma of the breast.
3. Negative for HER2-overexpression of the primary and/or metastatic tumour tissue detected by immunohistochemistry (DAKO 0-2) or genamplification detected by FISH.
4. Locally advanced or metastatic stage of disease not suitable for surgery or radiotherapy alone.
5. The following previous systemic treatment are eligible:

   adjuvant chemotherapy (except if capecitabine was included) adjuvant endocrine therapy palliative endocrine treatments treatment with bisphosphonates (adjuvant and/or palliative) treatment with immunotherapies (adjuvant and/or palliative)
6. Patients must have either measurable or nonmeasurable target lesions according to the WHO criteria (see Appendix 5).
7. At least 4 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside the radiation portal or there must be pathologic proof of progressive disease.
8. Complete radiology and tumor measurement work up within 4 weeks prior to registration.
9. Karnofsky performance status evaluation > or = 60%
10. Age >18 years
11. WBC > or = 3000 cells/microl, platelet count > or = 100,000 cells/microl.
12. Bilirubin < or = 2x the upper limit of normal for the institution (ULN); elevation of transaminases and alkaline phosphatase < 2.5x ULN or <5x ULN for patients with liver metastases.
13. Creatinine < or = 1,25 x upper normal value or creatinin-clearance > 50 ml/min (according to Cockroft Gault).
14. If of childbearing potential, negative pregnancy test. In addition the patient has to agree to use an effective method to avoid pregnancy for the duration of the study.
15. Female and male patients

Exclusion Criteria:

1. Known hypersensitivity reaction to the compounds or incorporated substances or known dihydropyrimidine dehydrogenase deficiency.
2. Concurrent immunotherapy or hormonal therapy (antihormonal, contraceptive and/or replacement therapy). Bisphosphonates may be continued.
3. Parenchymal brain metastases, unless adequately controlled by surgery and/or radiotherapy with complete resolution of symptoms and discontinuation of all steroids.
4. Life expectancy of less than 3 months.
5. Serious intercurrent medical or psychiatric illness that may interfere with the planned treatment (including AIDS and serious active infection).
6. History of other malignancy within the last 5 years which could affect the diagnosis or assessment of metastatic breast cancer.
7. Patients with indication for polychemotherapy.
8. Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
9. Treatment with sorivudine or derivates e.g. brivudin.
10. Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-07; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Any progression of disease or disease related death of a patient

SECONDARY OUTCOMES:
Any response (partial and complete) documented according to the WHO Criteria (s. App 6),
Time from complete or partial response until progression of disease or death due to any cause,
Any response (partial and complete) and stable disease of > 24 weeks duration documented according to the WHO Criteria (App. 6),
Any grade III/IV toxicity (NCI-CTC Version 2.0),
Premature treatment discontinuation,
Any dose reduction due to toxicity,
Any death of a patient,
EORTC QoL and modified Brunner Score,

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Kaufmann, MD, Principal Investigator — Klinikum der J. W. Goethe Universität, Universitätsfrauenklinik
Locations (1):
- J. W. Goethe Universität, Frauenklinik, Frankfurt am Main, Hesse, Germany

REFERENCES:
- See also: Click here for more information about this study: MoniCa Study — http://www.germanbreastgroup.de